CLINICAL TRIAL: NCT06026150
Title: Anatomical Variation of Femoral Nerve Location in Relation to Femoral Artery - An Ultrasonographic Evaluation
Brief Title: Anatomical Variations of Femoral Nerve Location in Relation to Femoral Artery
Status: Completed | Type: Observational
Sponsor: Rashid Hospital (Other Government)
Responsible Party: Principal Investigator, Kurian Palavilayil Thomas Vaidyan, Senior Specialist, Dept of Anesthesiology, Rashid Hospital
Other Study IDs: DSREC-06/2016_03
Record Dates: First submitted 2023-08-07; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Femoral Fractures
Keywords: femoral fracture; Ultrasound anatomy of femoral nerve
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasound scanning of inguinal area for femoral nerve and artery — ultrasound scanning of inguinal region is done in femoral fracture patient to identify femoral artery and nerve

SUMMARY:
The goal of this observational study is to learn about the relative position of femoral nerve in relation to the femoral artery in patients scheduled for femoral fractures using ultrasound scanning.

The classical description of femoral nerve is that it lies immediately near to artery, but it is not always true. The nerve lies at a varying distance from the artery.

The main question it aims to answer are:

• Is the age sex and Body Mass Index affect the relationship between femoral artery and nerve?

DETAILED DESCRIPTION:
The femoral nerve block is ideal for surgeries of the femur, knee, or anterior thigh and is often combined with a sciatic nerve block for near complete lower extremity analgesia. The classic teaching is that the femoral nerve lies lateral to femoral artery sandwiched between the fascia iliaca and iliopsoas muscle1.

Aim:

The objective of the study is to find out the anatomical variation in the site of the femoral nerve in relation to the femoral artery, with respect to the age, sex, weight and ethnicity of the patient.

ELIGIBILITY:
Inclusion Criteria:

* above the age of 18 coming for fixation of femoral fracture

Exclusion Criteria:

* below the age of 18
* patient not willing to participate
* patients with neurological illness that hinders from giving a valid consent
* patients with local pathology at inguinal region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: femoral fracture patients admitted in Rashid hospital and trauma centre Dubai
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-04-10 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Variability of anatomical position of Femoral Nerve with respect to Femoral artery - effect of age, sex and BMI | From the time the patient is positioned for ultrasound scanning to obtain a clear image of the femoral nerve until the measurement of the distance between the femoral nerve and artery is completed, assessed over a period of up to 6 hours.
  After positioning the patients with femoral fracture, ultrasound scanning of femoral nerve is done and the femoral nerve and arteries are identified. The distance between the femoral artery and nerve are measured using ultrasound.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fanara B, Christophe JL, Boillot A, Tatu L, Jochum D, Henri Y, Berthier F, Samain E. Ultrasound guidance of needle tip position for femoral nerve blockade: an observational study. Eur J Anaesthesiol. 2014 Jan;31(1):23-9. doi: 10.1097/01.EJA.0000435016.83813.aa. PMID 24145804
- [Background] Fingerman M, Benonis JG, Martin G. A practical guide to commonly performed ultrasound-guided peripheral-nerve blocks. Curr Opin Anaesthesiol. 2009 Oct;22(5):600-7. doi: 10.1097/ACO.0b013e32832f7643. PMID 19606024
- [Background] Baker MD, Gullett JP. Ultrasound-Guided Femoral Nerve Blocks. Pediatr Emerg Care. 2015 Dec;31(12):864-8; quiz 869-71. doi: 10.1097/PEC.0000000000000634. PMID 26626896
- [Background] Szucs S, Morau D, Iohom G. Femoral nerve blockade. Med Ultrason. 2010 Jun;12(2):139-44. PMID 21173942
- See also: Andrew T. Gray, Adam B. Collins, Ingeborg Schafhalter-Zoppoth, An introduction to femoral nerve and associated lumbar plexus nerve blocks under ultrasonic guidance, Techniques in Regional Anesthesia and Pain Management, Volume 8, Issue 4, 2004, Pages 155 — https://doi.org/10.1053/j.trap.2004.10.004

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT06026150/Prot_SAP_000.pdf